CLINICAL TRIAL: NCT01540851
Title: Adding Value in Knee Arthroplasty Post TKR Care Navigator Trial
Brief Title: Adding Value in Knee Arthroplasty Post-total Knee Replacement (TKR) Care Navigator Trial
Acronym: AViKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elena Losina, PhD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010p002597
Record Dates: First submitted 2012-02-21; First posted 2012-02-29 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-01

CONDITIONS: Osteoarthritis; Degenerative Joint Disease
Keywords: Osteoarthritis; Total Knee Replacement; total Knee Arthroplasty; Post operative recovery, TKA; Post-operative recovery TKR; Care Navigator
MeSH Terms: conditions — Osteoarthritis; Joint Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care Navigator Intervention Group (Active Comparator): Subjects randomized to the Care Navigator Intervention group will receive up to 10 telephone calls from a care navigator for 5 months post-operatively
  Interventions: Behavioral: Care Navigator
- Usual Care Group (Active Comparator): Subjects in the Usual Care group receive the current standard post-operative TKA care
  Interventions: Other: Standard Post-Operative TKA Care

INTERVENTIONS:
Behavioral: Care Navigator — Subjects assigned to the Care Navigator intervention group will receive 10 calls from a care navigator after discharge from the hospital for 5 months after their total knee replacement.
  Arms: Care Navigator Intervention Group
Other: Standard Post-Operative TKA Care — Subjects assigned to the Standard Post-Operative TKA Care group will receive the current standard of care for post-operative care
  Arms: Usual Care Group

SUMMARY:
The objectives of this research are to:

Conduct a proof of concept randomized controlled trial with up to 300 patients undergoing primary total knee replacement (TKA) at Brigham and Women's Hospital (BWH). The trial will compare a "Care Navigator" post-discharge intervention versus "Usual Care" post discharge management of patients undergoing TKA. The intervention will focus on the challenging process of transitions from the acute care hospital to inpatient or outpatient rehabilitation, and from inpatient rehabilitation to home.

The principal goals of the trial are:

1. To establish whether "Care Navigator" intervention improves functional outcomes as compared with the "Usual Care" treatment six months after TKA surgery.
2. To establish whether "Care Navigator" intervention is cost effective six months after TKA surgery.

The investigators hypothesize that:

1. Incorporating the Care Navigator role into the "Usual Care" treatment will increase TKA patients' rate of adherence to the rehabilitation protocol and improve functional outcomes.
2. Addition of a Care Navigator is cost-effective.

DETAILED DESCRIPTION:
The "Post-TKA Care Navigator" proof of concept intervention will be implemented as a randomized controlled trial. The investigators aim to identify and enroll a cohort of up to 300 subjects who have decided to undergo total knee replacement (TKA) at BWH. Subjects will be patients of the five orthopedic surgeons at Brigham and Women's Hospital who perform the most TKAs: Drs. Wright, Brick, Ready, Martin and Thornhill. Subjects will be followed from about two weeks prior to the operation to six months after discharge.

The investigators will assign patients into two groups, at random: 1) receiving current standard of post-operative care and 2) adding "Post-TKA Care Navigator". The role of the Care Navigator will be to follow up with patients via frequent telephone conversations, ranging from weekly during the first month to bi-weekly for the next 6 weeks to monthly by the 14th week post op. subjects assigned to the care navigator will receive up to 10 telephone calls over a period of 5 months. The goal of the Care Navigator would be to ensure or encourage compliance with physical therapy, triage patient concerns, questions and complaints, and identify those patients that require a call from a clinician to address a problem in the recovery process. For those issues that can be resolved easily at home the navigator would suggest strategies. The value of the post-TKA Care Navigator will be assessed by comparing functional status, satisfaction with surgery, utilization of health care, adherence to physical therapy, range of knee motion and intervention costs across the two randomized groups.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo primary TKA at Brigham & Women's Hospital
* Osteoarthritis is the principal underlying diagnosis
* Age >=40 at the projected date of TKA
* English-speaking

Exclusion Criteria:

* Osteoarthritis is not the principal underlying diagnosis (e.g. inflammatory arthritis)
* Dementia
* Psychological issues that preclude participation, as identified by participating surgeons
* Non-English speaker
* Diagnosis other than Osteoarthritis or secondary Osteoarthritis
* Age < 40 at the projected date of TKA
* Lives in a nursing home
* Implantation of Unicompartamental Knee Arthroscopy or Interpositional Arthroplasty
* Bilateral TKA in same admission (simultaneous)or planned bilateral within 6 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2011-07-24 (Actual); Primary Completion 2014-05-10 (Actual); Study Completion 2014-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Losina, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Losina E, Collins JE, Daigle ME, Donnell-Fink LA, Prokopetz JJ, Strnad D, Lerner V, Rome BN, Ghazinouri R, Skoniecki DJ, Katz JN, Wright J. The AViKA (Adding Value in Knee Arthroplasty) postoperative care navigation trial: rationale and design features. BMC Musculoskelet Disord. 2013 Oct 12;14:290. doi: 10.1186/1471-2474-14-290. PMID 24119081
- [Result] Losina E, Collins JE, Wright J, Daigle ME, Donnell-Fink LA, Strnad D, Usiskin IM, Yang HY, Lerner V, Katz JN. Postoperative Care Navigation for Total Knee Arthroplasty Patients: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2016 Sep;68(9):1252-9. doi: 10.1002/acr.22829. Epub 2016 Jul 28. PMID 26714179

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a tertiary academic medical center in Boston, MA
Groups:
- Care Navigator Intervention Group: Subjects randomized to the Care Navigator Intervention group will receive up to 10 telephone calls from a care navigator for 5 months post-operatively
  Care Navigator: Subjects assigned to the Care Navigator intervention group will receive 10 calls from a care navigator after discharged from the hospital for 5 months after their total knee replacement.
  Subjects assigned to the usual Care group will receive current standard of post-operative care
- Usual Care Group: Subjects in the Usual Care group receive the current standard post-operative TKA care
  Care Navigator: Subjects assigned to the Care Navigator intervention group will receive 10 calls from a care navigator after discharged from the hospital for 5 months after their total knee replacement.
  Subjects assigned to the usual Care group will receive current standard of post-operative care
Period: Overall Study
Arm/Group | Care Navigator Intervention Group | Usual Care Group
Started | 154 | 154
Completed | 133 | 136
Not Completed | 21 | 18
Not completed — Lost to Follow-up | 14 | 15
Not completed — Withdrawal by Subject | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Care Navigator Intervention Group | Usual Care Group | Total
Number analyzed (Participants) | 154 | 154 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8) | 67 (8) | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 93 | 186
  Male | 61 | 61 | 122
Region of Enrollment [Number; unit: participants]
  United States | 154 | 154 | 308
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31 (6) | 31 (6) | 31 (6)
WOMAC Physical Function score [Mean (Standard Deviation); unit: units on a scale] — The WOMAC Physical Function scale is scaled from 0 to 100, with 100 worst
  units on a scale | 42 (16) | 41 (19) | 41 (17)
WOMAC Pain score [Mean (Standard Deviation); unit: units on a scale] — The WOMAC Pain scale is scaled from 0 to 100, with 100 worst
  units on a scale | 42 (16) | 40 (19) | 41 (18)

OUTCOME MEASURES:

1. Primary Outcome: Change in WOMAC Physical Function
Description: The change in functional status will be measured using the WOMAC Physical Function scale at Baseline and 6 months
Time Frame: Change in functional status from baseline to 6 months
Population: The WOMAC Physical Function scale is scaled from 0 to 100, with 100 worst. Change in function was calculated as the WOMAC Physical Function score at 6 months minus the WOMAC Physical Function score at baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Care Navigator Intervention Group | Usual Care Group
Number analyzed (Participants) | 133 | 136
units on a scale | -30 [-33 to -27] | -27 [-30 to -23]

2. Secondary Outcome: Satisfaction
Description: Percentage of patients in each study arm who reported being very satisfied with the results of TKA
Time Frame: Measured at 6 months post TKA
Population: The proportion of participants who reported being very satisfied with the results of TKA was assessed using a 5-item Likert scale on the 6 month follow-up questionnaire
Measure: Number; unit: percentage of participants
Arm/Group | Care Navigator Intervention Group | Usual Care Group
Number analyzed (Participants) | 133 | 136
percentage of participants | 80 | 72

3. Secondary Outcome: Range of Motion
Description: Percentage of participants able to bend knee at least 120 degrees
Time Frame: 6 months after TKA
Population: Percentage of participants who self-reported on their 6 month questionnaire that they were able to bend their index knee to greater than 120 degrees
Measure: Number; unit: percentage of participants
Arm/Group | Care Navigator Intervention Group | Usual Care Group
Number analyzed (Participants) | 133 | 136
percentage of participants | 70 | 72

ADVERSE EVENTS:
Arm/Group | Care Navigator Intervention Group | Usual Care Group
Serious Adverse Events (participants affected / at risk) | 0/154 | 1/154
Other Adverse Events (participants affected / at risk) | 0/154 | 0/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Care Navigator Intervention Group (N=154) | Usual Care Group (N=154)
Death (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes